CLINICAL TRIAL: NCT06662149
Title: Dining Out in NYC: Using VR to Investigate the Influence of Multisensory Urban Design Factors on Eating Behavior in Emerging Adults
Brief Title: Exploring the Influence of Sensory Cues on Eating Behavior Using Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Travis Masterson, Assistant Professor and Director of the Health, Ingestive Behavior, and Technology Lab, Penn State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY00025849
Record Dates: First submitted 2024-10-22; First posted 2024-10-28 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Virtual Reality; Eating behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pleasant First (Experimental): Participants will experience the pleasant smell in the participant's first visit and the unpleasant smell in the participant's second visit.
  Interventions: Other: Pleasant Smell; Other: Unpleasant Smell
- Unpleasant First (Experimental): Participants will experience the unpleasant smell in the participant's first visit and the pleasant smell in the participant's second visit.
  Interventions: Other: Pleasant Smell; Other: Unpleasant Smell

INTERVENTIONS:
Other: Pleasant Smell — The participants will be in an environment with an assumed pleasant smell while consuming the meal.
Other: Unpleasant Smell — Participants will be in an environment with an assumed unpleasant smell while consuming the meal.

SUMMARY:
Many factors influence eating choices among humans (mood, taste, convenience, time of day, etc.). Finding simple ways to decrease food intake or improve food choices could improve weight status and overall health of the general population. The purpose of this study is to see if city and/or nature smells affect human eating behavior within a virtual reality-simulated outdoor café. The researchers of this study believe that a better understanding of how smells affect eating behavior could lead to public guidelines that direct the construction and layout of such outdoor eating environments to better support healthy behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-29
* Fluent in English
* Free of self-reported food allergies/food sensitivities
* No diagnosis of cognitive or physical disabilities/disorders that may affect appetite or eating behaviors (Examples include Major Depressive Disorder, dementia, or eating disorders)
* No diagnosis of disabilities that may affect sensory proprioception related to virtual reality (Examples include vertigo, epilepsy, and ataxia)
* Not color blind
* Does not experience anosmia (inability or weak ability to smell)
* Must have hair ≥3 cm in length at the cortisol sample site (roughly midline of the skull left to right and two inches up from the base of the hairline at the neck).
* No hair transplant in the last 6 months

Exclusion Criteria:

* Are younger than 18 or older than 29 years of age
* Not fluent in English
* Have self-reported food allergies
* Have a diagnosis of cognitive or physical disabilities that may affect appetite or eating behaviors (Examples include Major Depressive Disorder, dementia, or eating disorders)
* Have a diagnosis of disabilities that may affect sensory proprioception related to virtual reality (Examples include vertigo, epilepsy, and ataxia)
* Suffers from color blindness
* Suffers from anosmia (inability or weak ability to smell)
* Hair shorter than 3 cm in length at the cortisol sample site (roughly midline of the skull left to right and two inches up from the base of the hairline at the neck)
* Has had a hair transplant in the last 6 months

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Food Intake Day 1 | Measured once 5-10 minutes after the end of meal consumption
  Total weight of the meal and individual components of the meal are measured in grams before and after participant consumption. The difference is recorded as the amount consumed by the participant. Grams of food will be converted into kilocalories and reported as energy consumed as well.
Food Intake Day 2 | Measured 5-10 minutes after the end of meal consumption
  Total weight of the meal and individual components of the meal are measured in grams before and after participant consumption. The difference is recorded as the amount consumed by the participant. Grams of food will be converted into kilocalories and reported as energy consumed as well.
Scent Experience Questionnaire (SEQ) Baseline Visit 1 | Measured 5-10 minutes prior to entering VR environment at Visit 1
  Answered on a tablet; Participants respond to questions 1-3 using a visual analog scale with opposite descriptors on each end. Question 4 is open response that will be coded as a positive memory/scent or negative memory/scent.
  1. How pleasant or unpleasant is the smell you are experiencing? (low anchor: extremely unpleasant, high anchor: extremely pleasant)
  2. How intense is the smell you are experiencing? (low anchor: not detectable, high anchor: very strong)
  3. How familiar is the smell you are experiencing? (low anchor: completely unknown, high anchor: extremely familiar)
  4. Does the smell you are experiencing remind you of anything? If so, what?
Scent Experience Questionnaire (SEQ) Baseline Visit 2 | Measured 5-10 minutes prior to entering VR environment at Visit 2
  Answered on a tablet; Participants respond to questions 1-3 using a visual analog scale with opposite descriptors on each end. Question 4 is open response that will be coded as a positive memory/scent or negative memory/scent.
  1. How pleasant or unpleasant is the smell you are experiencing? (low anchor: extremely unpleasant, high anchor: extremely pleasant)
  2. How intense is the smell you are experiencing? (low anchor: not detectable, high anchor: very strong)
  3. How familiar is the smell you are experiencing? (low anchor: completely unknown, high anchor: extremely familiar)
  4. Does the smell you are experiencing remind you of anything? If so, what?
Scent Experience Questionnaire (SEQ) Post-VR Visit 1 | Measured 1-5 minutes after entering VR environment at Visit 1
  Answered on a tablet; Participants respond to questions 1-3 using a visual analog scale with opposite descriptors on each end. Question 4 is open response that will be coded as a positive memory/scent or negative memory/scent.
  1. How pleasant or unpleasant is the smell you are experiencing? (low anchor: extremely unpleasant, high anchor: extremely pleasant)
  2. How intense is the smell you are experiencing? (low anchor: not detectable, high anchor: very strong)
  3. How familiar is the smell you are experiencing? (low anchor: completely unknown, high anchor: extremely familiar)
  4. Does the smell you are experiencing remind you of anything? If so, what?
Scent Experience Questionnaire (SEQ) Post-VR Visit 2 | Measured 1-5 minutes after entering VR environment at Visit 2
  Answered on a tablet; Participants respond to questions 1-3 using a visual analog scale with opposite descriptors on each end. Question 4 is open response that will be coded as a positive memory/scent or negative memory/scent.
  1. How pleasant or unpleasant is the smell you are experiencing? (low anchor: extremely unpleasant, high anchor: extremely pleasant)
  2. How intense is the smell you are experiencing? (low anchor: not detectable, high anchor: very strong)
  3. How familiar is the smell you are experiencing? (low anchor: completely unknown, high anchor: extremely familiar)
  4. Does the smell you are experiencing remind you of anything? If so, what?

SECONDARY OUTCOMES:
Pleasure-Arousal-Dominance (PAD) Survey Baseline Visit 1 | Measured 5-10 minutes prior to entering VR environment at Visit 1
  Survey answered on a tablet; participant rates the following questions on a 1-9 scale, with 9 being a stronger feeling of the stated emotion.
  1. How would you rate the level of pleasure you are experiencing currently?
  2. How would you rate your current level of arousal (a state of excitement linked to an emotion)? 3 How would you rate the extent to which the emotion makes you feel you are in control of the situation?
Pleasure-Arousal-Dominance (PAD) Survey Baseline Visit 2 | Measured 5-10 minutes prior to entering VR environment at Visit 2
  Survey answered on a tablet; participant rates the following questions on a 1-9 scale, with 9 being a stronger feeling of the stated emotion.
  1. How would you rate the level of pleasure you are experiencing currently?
  2. How would you rate your current level of arousal (a state of excitement linked to an emotion)? 3 How would you rate the extent to which the emotion makes you feel you are in control of the situation?
Pleasure-Arousal-Dominance (PAD) Survey Post VR Visit 1 | Measured 1-5 minutes after entering VR environment at Visit 1
  Survey answered on a tablet; Participant is prompted with the following input: Imagine you are in the space you saw when wearing the headset. You are there after a long day's work. Now, how does the architectural space in the image make you feel?
  Scale of 1-9. A higher score indicates a stronger feeling in that dimension.
  1. How would you rate the level of pleasure you experienced in this space?
  2. How would you rate the level of arousal (a state of excitement linked to an emotion) you experienced in this space? 3 How would you rate the extent to which the emotion makes you feel you are in control of the situation?
Pleasure-Arousal-Dominance (PAD) Survey Post VR Visit 2 | Measured 1-5 minutes after entering VR environment at Visit 2
  Survey answered on a tablet; Participant is prompted with the following input: Imagine you are in the space you saw when wearing the headset. You are there after a long day's work. Now, how does the architectural space in the image make you feel?
  Scale of 1-9. A higher score indicates a stronger feeling in that dimension.
  1. How would you rate the level of pleasure you experienced in this space?
  2. How would you rate the level of arousal (a state of excitement linked to an emotion) you experienced in this space? 3 How would you rate the extent to which the emotion makes you feel you are in control of the situation?
Positive Affect Negative Affect Survey (PANAS) Baseline Visit 1 | Measured 5-10 minutes prior to entering VR environment at Visit 1
  Survey is taken on a tablet; Participant responds according to how much they are feeling that emotion at that moment with a 1-5 scale (1 is not at all and 5 is extremely).
  1. Interested
  2. Distressed
  3. Excited
  4. Upset
  5. Strong
  6. Guilty
  7. Scared
  8. Hostile
  9. Enthusiastic
  10. Proud
  11. Irritable
  12. Alert
  13. Ashamed
  14. Inspired
  15. Nervous
  16. Determined
  17. Attentive
  18. Jittery
  19. Active
  20. Afraid
Positive Affect Negative Affect Survey (PANAS) Baseline Visit 2 | Measured 5-10 minutes prior to entering VR environment at Visit 2
  Survey is taken on a tablet; Participant responds according to how much they are feeling that emotion at that moment with a 1-5 scale (1 is not at all and 5 is extremely).
  1. Interested
  2. Distressed
  3. Excited
  4. Upset
  5. Strong
  6. Guilty
  7. Scared
  8. Hostile
  9. Enthusiastic
  10. Proud
  11. Irritable
  12. Alert
  13. Ashamed
  14. Inspired
  15. Nervous
  16. Determined
  17. Attentive
  18. Jittery
  19. Active
  20. Afraid
Positive Affect Negative Affect Survey (PANAS) Post-VR Visit 1 | Measured 1-5 minutes after entering VR environment at Visit 1
  Survey is taken on a tablet; Participant responds according to how much they are feeling that emotion in response to the VR space with a 1-5 scale (1 is not at all and 5 is extremely).
  1. Interested
  2. Distressed
  3. Excited
  4. Upset
  5. Strong
  6. Guilty
  7. Scared
  8. Hostile
  9. Enthusiastic
  10. Proud
  11. Irritable
  12. Alert
  13. Ashamed
  14. Inspired
  15. Nervous
  16. Determined
  17. Attentive
  18. Jittery
  19. Active
  20. Afraid
Positive Affect Negative Affect Survey (PANAS) Post-VR Visit 2 | Measured 1-5 minutes after entering VR environment at Visit 2
  Survey is taken on a tablet; Participant responds according to how much they are feeling that emotion in response to the VR space with a 1-5 scale (1 is not at all and 5 is extremely).
  1. Interested
  2. Distressed
  3. Excited
  4. Upset
  5. Strong
  6. Guilty
  7. Scared
  8. Hostile
  9. Enthusiastic
  10. Proud
  11. Irritable
  12. Alert
  13. Ashamed
  14. Inspired
  15. Nervous
  16. Determined
  17. Attentive
  18. Jittery
  19. Active
  20. Afraid
State Anxiety Inventory (SAI) Baseline Visit 1 | Measured 5-10 minutes prior to entering VR environment at Visit 1
  Answered on a tablet; Read each statement and select the appropriate response to indicate how you feel right now, that is, at this very moment. Do not spend too much time on any one statement, but give the answer which seems to describe your present feelings best.
  Answered on a 1-4 scale:
  1 Not at all 2 A little 3 Somewhat 4 Very Much So
  1. I feel calm
  2. I feel secure
  3. I feel tense
  4. I feel strained
  5. I feel at ease
  6. I feel upset
  7. I am presently worrying over possible misfortunes
  8. I feel satisfied
  9. I feel frightened
  10. I feel uncomfortable
  11. I feel self confident
  12. I feel nervous
  13. I feel jittery
  14. I feel indecisive
  15. I am relaxed
  16. I feel content
  17. I am worried
  18. I feel confused
  19. I feel steady
  20. I feel pleasant
State Anxiety Inventory (SAI) Baseline Visit 2 | Measured 5-10 minutes prior to entering VR environment at Visit 2
  Answered on a tablet; Read each statement and select the appropriate response to indicate how you feel right now, that is, at this very moment. Do not spend too much time on any one statement, but give the answer which seems to describe your present feelings best.
  Answered on a 1-4 scale:
  1 Not at all 2 A little 3 Somewhat 4 Very Much So
  1. I feel calm
  2. I feel secure
  3. I feel tense
  4. I feel strained
  5. I feel at ease
  6. I feel upset
  7. I am presently worrying over possible misfortunes
  8. I feel satisfied
  9. I feel frightened
  10. I feel uncomfortable
  11. I feel self confident
  12. I feel nervous
  13. I feel jittery
  14. I feel indecisive
  15. I am relaxed
  16. I feel content
  17. I am worried
  18. I feel confused
  19. I feel steady
  20. I feel pleasant
State Anxiety Inventory (SAI) Post-VR Visit 1 | Measured 1-5 minutes after entering VR environment at Visit 1
  Answered on a tablet; Read each statement and select the appropriate response to indicate how you feel right now, that is, at this very moment. Do not spend too much time on any one statement, but give the answer which seems to describe your present feelings best.
  Answered on a 1-4 scale:
  1 Not at all 2 A little 3 Somewhat 4 Very Much So
  1. I feel calm
  2. I feel secure
  3. I feel tense
  4. I feel strained
  5. I feel at ease
  6. I feel upset
  7. I am presently worrying over possible misfortunes
  8. I feel satisfied
  9. I feel frightened
  10. I feel uncomfortable
  11. I feel self confident
  12. I feel nervous
  13. I feel jittery
  14. I feel indecisive
  15. I am relaxed
  16. I feel content
  17. I am worried
  18. I feel confused
  19. I feel steady
  20. I feel pleasant
State Anxiety Inventory (SAI) Post-VR Visit 2 | Measured 1-5 minutes after entering VR environment at Visit 2
  Answered on a tablet; Read each statement and select the appropriate response to indicate how you feel right now, that is, at this very moment. Do not spend too much time on any one statement, but give the answer which seems to describe your present feelings best.
  Answered on a 1-4 scale:
  1 Not at all 2 A little 3 Somewhat 4 Very Much So
  1. I feel calm
  2. I feel secure
  3. I feel tense
  4. I feel strained
  5. I feel at ease
  6. I feel upset
  7. I am presently worrying over possible misfortunes
  8. I feel satisfied
  9. I feel frightened
  10. I feel uncomfortable
  11. I feel self confident
  12. I feel nervous
  13. I feel jittery
  14. I feel indecisive
  15. I am relaxed
  16. I feel content
  17. I am worried
  18. I feel confused
  19. I feel steady
  20. I feel pleasant
Affect and Spatial Experience Scale (ASE) | Measured 5-10 minutes after the end of meal consumption and VR experience at visit 1
  Answered on a tablet; Participants rate their experience with the virtual reality environment on a -10 to 10 scale with opposite descriptors on either end of the scale and 10 being the most like the stated attribute
  1. Pleasantness: unpleasant vs. pleasant
  2. Liveliness: Lifeless vs. lively
  3. Beauty: ugly vs. beautiful
  4. Familiarity: Unfamiliar vs. familiar
  5. Excitement: not exciting vs. exciting
  6. Novelty: Traditional vs. novel
  7. Spaciousness: narrow vs. spacious
  8. Simplicity: Complex vs. simple
  9. Enclosure: Open vs. closed
  10. Order: Chaotic vs. ordered
  11. Lightness: Overwhelming vs. light
  12. Harmony: Not harmonious vs. harmonious
  13. Calmness: Stressful vs. calming
  14. Warmth: Cold vs. warm
  15. Brightness: Dark vs. bright
  16. Experience: Bad vs. good
  17. Comfort: Uncomfortable vs. comfortable
  18. Naturalness: Artificial vs. natural
  19. Cheerfulness: Depressing vs. cheerful
  20. Symmetry: Asymmetrical vs. symmetrical
VR Presence Questionnaire Visit 1 | Measured once 5-10 minutes after the end of meal consumption and the VR experience at visit 1
  Answered on a tablet; participants marked on a visual analog scale from 0-100 how they felt in the VR with 0 being not at all and 100 being very much
  1. In the virtual world, I had a sense of "being there"
  2. I felt that the virtual world surrounded me.
  3. I felt like I was just perceiving pictures.
  4. I did not feel present in the virtual space.
  5. I had a sense of acting in the virtual space, rather than operating something from outside.
  6. I felt present in the virtual space.
  7. How aware were you of the real world surrounding while navigating in the virtual world? (i.e. sounds, room temperature, other people, etc.)?
  8. I was not aware of my real environment.
  9. I still paid attention to the real environment.
  10. I was completely captivated by the virtual world.
  11. How real did the virtual world seem to you?
  12. How much did your experience in the virtual environment seem consistent with your real world experience ?
VR Presence Questionnaire Visit 2 | Measured once 5-10 minutes after the end of meal consumption and the VR experience at visit 2
  Answered on a tablet; participants marked on a visual analog scale from 0-100 how they felt in the VR with 0 being not at all and 100 being very much
  1. In the virtual world, I had a sense of "being there"
  2. I felt that the virtual world surrounded me.
  3. I felt like I was just perceiving pictures.
  4. I did not feel present in the virtual space.
  5. I had a sense of acting in the virtual space, rather than operating something from outside.
  6. I felt present in the virtual space.
  7. How aware were you of the real world surrounding while navigating in the virtual world? (i.e. sounds, room temperature, other people, etc.)?
  8. I was not aware of my real environment.
  9. I still paid attention to the real environment.
  10. I was completely captivated by the virtual world.
  11. How real did the virtual world seem to you?
  12. How much did your experience in the virtual environment seem consistent with your real world experience ?
VR Preference Questionnaire Visit 1 | Measured once 5-10 minutes after the end of meal consumption and the VR experience at visit 1
  Answered on a tablet; Participants would rank on a 0-8 point scale: for question 1-None, a few minutes, half an hour, one hour, a few hours, a day, a few days, many many days; for questions 2-5-not at all, very slight, slight, slight to moderate, moderate, much, very much, extremely so
  1. How much time would you like to spend in the virtual environment?
  2. How much would you try to leave or get out of this place?
  3. How much would you enjoy exploring around?
  4. How much would you avoid any looking around or exploration of the space?
  5. How much would you choose to enter this eating environment?
VR Preference Questionnaire Visit 2 | Measured once 5-10 minutes after the end of meal consumption and the VR experience at visit 2
  Answered on a tablet; Participants would rank on a 0-8 point scale: for question 1-None, a few minutes, half an hour, one hour, a few hours, a day, a few days, many many days; for questions 2-5-not at all, very slight, slight, slight to moderate, moderate, much, very much, extremely so
  1. How much time would you like to spend in the virtual environment?
  2. How much would you try to leave or get out of this place?
  3. How much would you enjoy exploring around?
  4. How much would you avoid any looking around or exploration of the space?
  5. How much would you choose to enter this eating environment?
Hair Cortisol | Measured once 15 minutes prior to entering VR environment at Visit 1
  The 3-month concentration of cortisol in the participant's hair will be recorded in picograms per milligram--higher values mean higher stress over the past 3 months.

OTHER OUTCOMES:
Reasons Individuals Stop Eating Questionnaire | Measured once 5-10 minutes after the end of meal consumption and the VR experience at visit 2
  Answered on a tablet; participants rate on a scale from 1-7 how much each statement reflects their typical behavior
  Rating Scale
  1, Never | 2, Rarely | 3, Seldom | 4, Sometimes | 5, Often | 6, Usually | 7, Always
  Prompt participants receive: Think about eating a typical dinner meal in your home. For each statement below, identify the frequency that best reflects how often you experience this as a reason that you stop eating a typical dinner at home.
Adult Eating Behavior Questionnaire | Measured once 5-10 minutes after the end of meal consumption and the VR experience at visit 2
  Answered on a tablet; participants rate on a scale from 1-5 how much each statement reflects their typical behavior
  Rating Scale
  1, Strongly disagree | 2, Disagree | 3, Neither agree or disagree | 4, Agree | 5, Strongly agree
External Cue Reactivity Questionnaire | Measured once 5-10 minutes after the end of meal consumption and the VR experience at visit 2
  Answered on a tablet; participants rate on a scale from 1-4 how often the statement is true for them
  Rating Scale
  1, Rarely | 2, Sometimes | 3, Often | 4, A lot
  Questions:
  1. I want foods or drinks that I see others eating.
  2. I notice snack or drink vending machines.
  3. I want to eat when people talk about food.
  4. I notice restaurant signs/logos.
  5. I notice snacks at check-out aisles.
  6. I like certain snacks because of the packaging.
  7. I notice the sound of food cooking.
  8. I want to eat when I hear a snack being opened.
  9. I expect to snack when I'm in my car.
Three Factor Eating Questionnaire | Measured once 5-10 minutes after the end of meal consumption and the VR experience at visit 2
  Answered on a tablet; participants rate on a scale from 1-4 how true the statement is for them
  Rating Scale
  1, Definitely false | 2, Mostly false | 3, Mostly true | 4, Definitely true
Engagement Questionnaire | Measured once 5-10 minutes after the end of meal consumption and the VR experience at visit 2
  Answered on a tablet; participants rate on a scale from 1-7 how much they agree with each statement. Questions 1-3 were reverse scored.
  Rating Scale
  1, Strongly disagree | 2, Disagree | 3, Somewhat disagree | 4, Neutral | 5, Somewhat agree | 6, Agree | 7, Strongly agree
Visual Analog Scale of Hunger and Thirst Baseline Visit 1 | Measured 5-10 minutes prior to entering VR environment at Visit 1
  Answered on a tablet; Participants rate their hunger, thirst, fullness, and nausea on a 0-100 scale where 0 is not at all and 100 is extremely.
Visual Analog Scale of Hunger and Thirst Baseline Visit 2 | Measured 5-10 minutes prior to entering VR environment at Visit 2
  Answered on a tablet; Participants rate their hunger, thirst, fullness, and nausea on a 0-100 scale where 0 is not at all and 100 is extremely.
Visual Analog Scale of Hunger and Thirst Post Visit 2 | Measured 5-10 minutes after the end of meal consumption and VR experience at Visit 2
  Answered on a tablet; Participants rate their hunger, thirst, fullness, and nausea on a 0-100 scale where 0 is not at all and 100 is extremely.
Visual Analog Scale of Hunger and Thirst Post Visit 1 | Measured 5-10 minutes after the end of meal consumption and VR experience at Visit 1
  Answered on a tablet; Participants rate their hunger, thirst, fullness, and nausea on a 0-100 scale where 0 is not at all and 100 is extremely.

CONTACTS AND LOCATIONS:
Overall Officials: Travis Masterson, Principal Investigator — The Pennsylvania State University
Locations (1):
- Health, Ingestive Behavior, and Technology Laboratory of Pennsylvania State University, State College, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No